CLINICAL TRIAL: NCT04085029
Title: Role of Ablative Radiotherapy in the Management of Metastatic Disease: A Patient Data Registry
Status: Recruiting | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00103137
Record Dates: First submitted 2019-09-09; First posted 2019-09-11 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Oligometastasis; Metastatic Cancer
Keywords: Ablative radiotherapy
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to provide a registry of participants in order to assess the acute adverse event rates following ablative radiotherapy for metastatic disease.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years of age
* Radiographic evidence of metastatic disease (may include oligoprogression, oligorecurrence or oligometastasis) at the time of study enrollment
* Planned to receive, currently receiving, or have completed hypofractionated image guided radiotherapy (ablative radiotherapy) to an extracranial site(s)
* Patient must sign study-specific informed consent

Exclusion Criteria:

• None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients at Duke University Health System Radiation Oncology treatment facilities or Durham VA Medical Center
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2019-09-26 (Actual); Primary Completion 2029-09 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
Occurrence of acute adverse events following radiotherapy | 90 Days

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Salama, MD, Principal Investigator — Duke University
Locations (5):
- United States (5):
  - Duke Cancer Institute Cary, Cary, North Carolina
  - Durham Veterans Administration Health Care System (DVAHCS), Durham, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Duke Women's Cancer Care Raleigh, Raleigh, North Carolina
  - Duke Raleigh Hospital, Raleigh, North Carolina

IPD SHARING:
Plan to Share IPD: No